CLINICAL TRIAL: NCT06495333
Title: Fecal Microbiota Analysis of PNPLA3 Polymorphism in Hispanic Patients With Metabolic Dysfunction Associated Steatotic Liver Disease
Brief Title: Fecal Microbiota Analysis of PNPLA3 Polymorphism in Hispanic Patients With MASLD
Acronym: MPM
Status: Recruiting | Type: Observational
Sponsor: Fundacion de Investigacion Science and Education (Other)
Responsible Party: Sponsor
Other Study IDs: FDI-2024-001
Record Dates: First submitted 2024-05-31; First posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Metabolic Dysfunction-associated Steatotic Liver Disease
Keywords: MASLD; NAFLD
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — whole blood and fecal sample
Oversight: Data Monitoring Committee: No

SUMMARY:
Metabolic Dysfunction-Associated Steatotic Liver Disease (MASLD) is the most common cause of liver disease worldwide. The condition is defined by fat accumulation exceeding 5% of liver weight not explained by at-risk alcohol intake. Risk factors include obesity, diabetes, genetic variants, dietary factors, and gut microbiota alterations. However, the interdependence of these factors and their individual impact on disease severity remain unclear. The investigators aim to investigate the changes in the gut microbiome of Hispanics living in Puerto Rico with MASLD associated with wild-type and mutated genotype status of PNPLA3 rs738409, a strong genetic contributor to MASLD. In this cross-sectional study, blood and fecal samples will be collected from participants who have completed a non-invasive transient elastography test (FibroScan) to measure the extent of hepatic steatosis (fat in the liver). Genotyping for the PNPLA3 rs738409 variant will be conducted. Fecal samples will be collected to analyze the V4 region of the 16S rRNA gene for intestinal microbiota characterization. Alpha and beta diversity analysis will be measured by MASLD status and PNPLA3 genotype to evaluate biodiversity within and between samples.

DETAILED DESCRIPTION:
The liver is the powerhouse of the body, overseeing many functions such as the production of clotting factors, sugars, fats, and the metabolism of drugs. MASLD is the most common chronic liver disease worldwide, affecting one in three adults and one in ten children. MASLD, more commonly referred to as "fatty liver," can lead to fat accumulation in liver cells or steatosis and is strongly associated with obesity and diabetes. The disease is usually considered a silent condition with few symptoms until advanced liver disease or cirrhosis develops. Fortunately, fatty liver may be reversed by adopting a healthy lifestyle, including weight loss and exercise. However, the pathogenesis of MASLD remains incompletely understood, and the Hispanic subpopulation is affected the most.

A multi-hit model has been proposed that most accurately describes both the development of simple steatosis and its transition from simple steatosis to progressive stages of the disease. In this model, a close interaction between dietary, environmental, and genetic factors with insulin resistance, lipotoxicity, and fat metabolism comprises multiple insults acting together on predisposed subjects to induce MASLD. This model has led to the understanding that the interplay between diet, genetics, and gut microbiota is of utmost importance in the development and progression of the condition. As a multi-factorial disease, assigning specific disease pathways to the overall phenotype has been challenging. Still, it is important to investigate associations between its risk factors to direct therapeutic interventions to the most relevant pathways.

Looking at two of the most relevant risk factors, this study aims to investigate whether there are any differences in the taxonomic composition of the gut microbiota between Hispanic patients with MASLD with different PNPLA3 genotypes. The PNPLA3 (patatin-like phospholipase domain-containing protein 3) polymorphism has been implicated in the pathogenesis and progression of the condition. However, the role of PNPLA3 polymorphism in shaping the fecal microbiota composition in Hispanic patients with MASLD remains unclear. Once fecal and blood samples are collected from a cohort of Hispanic individuals with MASLD, fecal microbiota sequencing and PNPLA3 genotyping will be done. Findings will reveal whether there are significant alterations in the fecal microbiota composition in relation to PNPLA3 polymorphism in Hispanic patients with MASLD. Results could provide evidence for a potential link between PNPLA3 polymorphism and fecal microbiota composition in Hispanic individuals with MASLD.

ELIGIBILITY:
Inclusion Criteria:

A subject must meet the following criteria to be eligible for inclusion in the study:

Patient must be of Hispanic ethnicity residing in Puerto Rico. Age 21 to 75 years old at time of informed consent. Evidence of MASLD by vibration-controlled transient elastography (FibroScan) controlled attenuation parameter (CAP) (value must be greater than or equal to 248 dB/m).

Willing and able to provide informed consent signed by study subject. Willing and able to understand and complete study-related procedures.

Exclusion Criteria:

A subject who meets any of the following criteria will be excluded from the study:

Excessive alcohol intake for ≥3 months during past year prior to screening (>3 units/day for males and >2 units/day for female is generally considered excessive).

History of liver transplant, or current placement on a liver transplant list. History of viral and resolved hepatitis (Hepatitis B or C) or human immunodeficiency virus (HIV).

Use of antibiotics within 14 days of screening.

Ages: 21 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The aim of this study is to determine the changes in the gut microbiome in Hispanics living in Puerto Rico with MASLD associated to wild-type and mutated PNPLA3 genotype status will also be assessed in this study population. To maintain homogeneity of the study population and to achieve the study objectives, the study will only be including individuals who self-identify as Hispanic and currently reside in Puerto Rico. Exclusion of non-Hispanic individuals is necessary to ensure that obtained results are representative of the Hispanic population in Puerto Rico and can be generalized to this population.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-07-05 (Actual); Primary Completion 2024-12-28 (Estimated); Study Completion 2025-08-20 (Estimated)

PRIMARY OUTCOMES:
Microbiota characterization | 1 year
  To determine the changes in the gut microbiome of Hispanics living in Puerto Rico with MASLD associated to wild-type and mutated genotype status of PNPLA3 rs738409, a strong genetic contributor to MASLD.
Microbiota diversity based on eating patterns | 1 year
  To determine microbiome diversity in Hispanics with different eating patterns.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Pi, BS, Study Chair — FDI Clinical Research
Locations (1):
- FDI Clinical Research, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Buzzetti E, Pinzani M, Tsochatzis EA. The multiple-hit pathogenesis of non-alcoholic fatty liver disease (NAFLD). Metabolism. 2016 Aug;65(8):1038-48. doi: 10.1016/j.metabol.2015.12.012. Epub 2016 Jan 4. PMID 26823198
- [Background] Chan WK, Chuah KH, Rajaram RB, Lim LL, Ratnasingam J, Vethakkan SR. Metabolic Dysfunction-Associated Steatotic Liver Disease (MASLD): A State-of-the-Art Review. J Obes Metab Syndr. 2023 Sep 30;32(3):197-213. doi: 10.7570/jomes23052. Epub 2023 Sep 13. PMID 37700494
- [Background] Godoy-Matos AF, Silva Junior WS, Valerio CM. NAFLD as a continuum: from obesity to metabolic syndrome and diabetes. Diabetol Metab Syndr. 2020 Jul 14;12:60. doi: 10.1186/s13098-020-00570-y. eCollection 2020. PMID 32684985
- [Background] Lang S, Martin A, Zhang X, Farowski F, Wisplinghoff H, J G T Vehreschild M, Krawczyk M, Nowag A, Kretzschmar A, Scholz C, Kasper P, Roderburg C, Mohr R, Lammert F, Tacke F, Schnabl B, Goeser T, Steffen HM, Demir M. Combined analysis of gut microbiota, diet and PNPLA3 polymorphism in biopsy-proven non-alcoholic fatty liver disease. Liver Int. 2021 Jul;41(7):1576-1591. doi: 10.1111/liv.14899. Epub 2021 May 7. PMID 33896117
- [Background] Tilg H, Adolph TE, Moschen AR. Multiple Parallel Hits Hypothesis in Nonalcoholic Fatty Liver Disease: Revisited After a Decade. Hepatology. 2021 Feb;73(2):833-842. doi: 10.1002/hep.31518. Epub 2021 Feb 6. No abstract available. PMID 32780879
- [Background] Romeo S, Kozlitina J, Xing C, Pertsemlidis A, Cox D, Pennacchio LA, Boerwinkle E, Cohen JC, Hobbs HH. Genetic variation in PNPLA3 confers susceptibility to nonalcoholic fatty liver disease. Nat Genet. 2008 Dec;40(12):1461-5. doi: 10.1038/ng.257. Epub 2008 Sep 25. PMID 18820647
- See also: New MASLD Nomenclature — http://www.aasld.org/new-masld-nomenclature
- See also: Nonalcoholic Fatty Liver Disease (NAFLD) — https://www.liverfoundation.org/liver-diseases/fatty-liver-disease/nonalcoholic-fatty-liver-disease-nafld/
- See also: Fatty liver disease diet: What foods help prevent and reverse fatty liver?. — https://www.uchicagomedicine.org/forefront/gastrointestinal-articles/2021/september/fatty-liver-disease-diet
- See also: Non-Alcoholic Fatty Liver Disease: Assessment and Management. — https://www.ncbi.nlm.nih.gov/books/NBK384735/